CLINICAL TRIAL: NCT06836622
Title: Correlation Between the Values of Carotid-Femoral, Oscillometric and Estimated Pulse Wave Velocity
Brief Title: Carotid-Femoral, Oscillometric and Estimated Pulse Wave Velocity
Acronym: CF-O-E-PWV
Status: Enrolling by invitation | Type: Observational
Sponsor: Hospital de Base (Other)
Responsible Party: Principal Investigator, JOSE FERNANDO VILELA-MARTIN, PhD, Hospital de Base
Other Study IDs: cfPWV, brPWV and ePWV
Record Dates: First submitted 2025-02-06; First posted 2025-02-20 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Hypertension; Arterial Stiffness; Pulse Wave Analysis; Pulse Wave Velocity
Keywords: Arterial stiffness; Hypertension; Pulse wave velocity
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Adults older than eighteen with elevated office BP, treated and untreated.: All participants were referred by a physician to perform ambulatory blood pressure monitoring (ABPM) to confirm a hypertension diagnosis or evaluate uncontrolled hypertension.

SUMMARY:
What is the purpose of this research? This research aims to compare three different methods of measuring pulse wave velocity, which is the main parameter used for assessing arterial stiffness. This parameter is as important as blood pressure in predicting future cardiovascular risk.

The investigators intend to compare carotid-femoral pulse wave velocity, which is the gold standard for measuring arterial stiffness, with brachial pulse wave velocity measured using a device similar to a blood pressure monitor and a mathematical formula validated in a large European population.

Who is eligible for this survey? Anyone aged 18 or older who has been invited may participate, provided they sign an informed consent form.

Where will the field research be conducted? The research will be conducted at a health center specializing in the treatment of hypertension. This center is a reference for outpatient blood pressure monitoring in the city of Uberaba (MG), Brazil.

Which procedures will be performed by research participants? All participants who consent will answer some questions about their demographic and health information. A trained nurse will measure their weight, height, and blood pressure after a 5-minute rest, and then measure carotid-femoral pulse wave velocity. The participant will lie down on a bed and the nurse will place a sensor on the middle of their neck and the groin. The device will automatically deliver the parameters. At least three measurements are required for each participant. Measurements normally take between 10 and 15 minutes. Then, participants will wear a device to record blood pressure and pulse wave velocity for 24 hours. The nurse will fit the cuff around the participant's arm and attach the monitoring device to a belt around their waist. The device will take measurements every 20 to 30 minutes. 24 hours later, the participant must return to the research venue to have the equipment removed.

What are the risks and adverse events of the procedures? There are no known risks or adverse events (AEs) associated with carotid-femoral pulse wave velocity measurements. The risks of this research are minimal, limited to discomfort during the AMBP recording, which occurs at a low frequency. However, excessive arm pain, allergic reactions, and edema may occur. To minimize these risks, a nurse will be available via telephone to aid all participants during the AMBP recordings.

DETAILED DESCRIPTION:
•BACKGROUND It is estimated that 1 in 4 adults suffers from hypertension, including 40% of those over the age of 25. Blood pressure tends to be higher in older adults, and in developed countries, an estimated 9 in 10 adults who live to 80 years of age will develop hypertension. Over the decades, data have shown a positive and continued association between BP values and the occurrence of heart attacks and strokes.

Artery stiffening (AS) and increased pulsatile diameter were identified as standard features of hypertension in individuals aged between 40 and 50 years, and have emerged as two of the most valuable, distinctive, and independent predictors of cardiovascular events.

Considering that pulse waves from the aorta travel to the peripheral arterial vessels more quickly in stiffer vessels, some authors suggested, in 1987, that aortic pulse wave velocity (PWV) could give reliable information about arterial stiffness. In the last few decades, due to numerous studies demonstrating that carotid-femoral PWV (cf-PWV) is a strong independent predictor of total mortality and major cardiovascular (CV) events, PWV has become a gold standard biological marker of arterial stiffness.

Therefore, in medical literature, arterial stiffness has long been strongly associated with pulse wave velocity (PWV). PWV is calculated as the distance traveled by the arterial pulse between proximal and distal vascular sites by the corresponding time interval. Currently, invasive catheter-based PWV measurement is used only in validation studies due to its complexity, high cost, and ethical limitations. Over the last two decades, several noninvasive devices for measuring PWV have been validated in published studies.

Simultaneous carotid and femoral artery measurement is the non-invasive reference for studies involving cf-PWV. Two investigators should conduct the measurement, ensuring a minimum recording time of 10 cardiac cycles. Ideally, measurements should be performed at the same time; ECG-gated sequential measurements are the second-best alternative. The recordings from the right carotid and right femoral arteries are preferred. Transit time should be determined using the intersecting tangent method. Commercial devices that currently fulfill these criteria are the Complior Analyze device (Alam Medical, Saint Quentin Fallavier, France) and the original Sphygmocor system that used tonometry for both carotid and femoral pulse wave acquisitions (discontinued; ATCOR Medical, CardieX Pty, Ltd, Sydney, NSW, Australia).

In recent decades, new devices have enabled the measurement of PWV by recording signals at more peripheral areas using brachial cuffs. The Mobil-O-Graph is one of them. It is an automated oscillometric brachial cuff-based ambulatory BP monitoring device that can measure PWV (br-PWV) by proprietary algorithms. The br-PWV can independently predict mortality in chronic kidney disease (CKD) stage 2-4. It is also associated with an increased risk of cardiovascular events and all-cause mortality in hemodialysis patients.

Additionally, mathematical formulas can estimate PWV (ePWV) based on the Reference Values for Arterial Stiffness Collaboration, published nearly fifteen years ago. The aim of this publication was to define the determinants and reference values of cf-PWV. This study demonstrated age and BP accounted for PWV and its variance in a population. Therefore, the authors proposed two formulas that used mean BP and age to calculate cf-PWV.

Analyses of data from two European populations demonstrated that e-PWV was able to predict major cardiovascular events regardless of the Systematic COronary Risk Evaluation (SCORE), the Framingham risk score (FRS), and the cf-PWV. Another recent study found an association between ePWV and CV diseases and all-cause mortality in a Chinese population, independent of CV risk factors. In addition, ePWV predicted cardiovascular events and mortality in patients with suspected coronary artery disease, and it also improved risk stratification in hospitalized COVID-19 patients, beyond conventional risk factors and scores.

Therefore, since the Mobil-o-Graph device measures PWV using an algorithm based on age and BP values, it is an expensive option. In contrast, e-PWV estimates pulse wave velocity solely through mathematical formulas. This study aimed to evaluate the correlation between the ePWV and br-PWV with the gold standard cf-PWV.

• METHODS Population and Location Subjects were selected from a health center specializing in diagnosing and treating non-communicable diseases in the city of Uberaba, Brazil, who were referred to undergo ambulatory blood pressure monitoring (ABPM) to confirm a hypertension diagnosis or evaluate uncontrolled hypertension.

Data Collection Demographic and clinical data were collected from all subjects, including previous reports of acute myocardial infarction, acute coronary syndrome, coronary or other arterial revascularization, stroke, transient ischemic attack, aortic aneurysm, peripheral artery disease, and severe chronic kidney disease (CKD). They also had their weight, height, and waist circumference measured. A nursing assistant conducted BP measurements and pulse wave analyses (PWA).

Blood Pressure Measurement

The office BP (OBP) measurements followed recommended guidelines to ensure accurate pressure values. A nursing assistant operated a Microlife device model AFIB BPA200 (Onbo Electronic Co, Shenzhen, China). This device operates in Microlife Average Mode, which takes three consecutive measurements and calculates the average BP value. The nursing assistant took one set of three BP measurements.

Carotid-Femoral Pulse Wave Analyses

After having their BP measured, participants rested for 10 minutes in the supine position. The assistant then performed the pulse wave analyses (PWA) utilizing a Complior Analyze device (ALAM MEDICAL, Saint Quentin Fallavier, France). The determination of PWA followed all the standards set in the 2012 Expert Consensus Document for measuring Aortic Stiffness, including conducting procedures in a quiet room with stable temperature. The device uses non-invasive pressure sensors to record arterial pulse simultaneously. One sensor was positioned at the carotid artery site, and the other at the femoral artery site, on the dominant side of the body. Complior automatically calculated PWV as PWV =ΔL/ΔT, where ΔT represents the transit time and ΔL being the effective distance between the two recording sites. Transit time was measured using the intersecting tangent method, and the distance was estimated as 0.8× the measured carotid-femoral distance.

Brachial Pulse Wave Analyses

Finally, for data collection, all subjects recorded twenty-four hours of ABPM utilizing a Dyna-Mapa monitor (Cardios, São Paulo, Brazil), equipped with an appropriately-sized cuff on their non-dominant arm. The device was set up to take both BP and br-PWV readings every 20 minutes throughout the day (7 AM to 11 PM). During the night (11 PM to 7 AM), BP was measured every 30 minutes, and br-PWV was measured hourly. For ABPM analyses, 'night' was defined as the period between going to bed and waking up. All recommended protocols were strictly followed in order to ensure quality recordings.

Calculation of Estimated Pulse Wave Velocity To determine the appropriate equation for calculating ePWV, we assessed the prevalence of healthy and at-risk individuals in the sample population. Healthy individuals were those who presented no risk factors and a non-elevated BP (< 140 and 90 mmHg). On the other hand, the at-risk group included individuals with elevated BP (>140 or 90 mmHg) or at least one risk factor, such as history of hypertension, dyslipidemia, diabetes, smoking, obesity (BMI ≥ 30 kg/m2), abdominal waist circumference at risk (> 102 cm in males, > 88 cm in females). Therefore, we calculated e-PWV using equations 1 and 2, derived from the Reference Values for Arterial Stiffness Collaboration, based on age and MBP, as follows.

At-risk individuals: e-PWV = 9.58748315543126-0.402467539733184*age+4.56020798207263*10-3*age2-2.6207705511664*10-5*age2*MBP+3.1762450559276*10-3*age*MBP-1.832150382185*10-2*MBP.

Healthy individuals: e-PWV = 4.62 - 0.13*age + 0.0018*age^2 + 0.0006*age*MBP + 0.0284*MBP We used the average of the first three BP measurements to estimate MBP, which was calculated as 40% of office pulse pressure plus diastolic BP; MBP = diastolic BP+ 0.4*(systolic BP- diastolic BP).

Statistical Analysis

The normal distribution of the variables will be analyzed. Depending on the results, data will be expressed through proportions, mean, or median. We will apply the chi-squared test to compare proportions. If the distribution is normal, we will use the concordance correlation coefficient (Pc) to assess the association, precision (p), and accuracy among cf-PWV, br-PWV, and e-PWV. If the distribution is abnormal, we will use the Rank correlation to assess the relationship among all PWV metrics. Additionally, we will use a Bland-Altman plot to investigate the agreement among cf-PWV, br-PWV, and e-PWV values.

The databases will be built using Microsoft Excel, and the statistical analyses will be conducted using MedCalc. All participants will provide written informed consent to participate in the study.

ELIGIBILITY:
Inclusion Criteria :

- Individuals older than 18 with an elevated office blood pressure :

* suspected hypertension diagnosis or
* uncontrolled hypertension under treatment

Exclusion Criteria:

24-hour ABPM recordings presenting:

* less than 70% of the expected measurements or
* fewer than 20 valid awake or seven valid sleeping measurements or
* fewer than two valid daytime and one valid night-time measurement per hour

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals older than 18 with a suspected hypertension diagnosis or under treatment who were referred to record twenty-four hours of ABPM either to confirm a hypertension diagnosis or evaluate uncontrolled hypertension. The participants will be selected in a specialized center in inner Brazil to diagnose and treat non-communicable diseases.
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-03-02 (Estimated)

PRIMARY OUTCOMES:
Concordance correlation coefficient | Through study completion, an average of 1 year.
  The concordance correlation coefficient evaluates the degree to which pairs of observations fall on the 45° line through the origin. The concordance correlation coefficient (ρc) contains a measurement of precision (ρ) and accuracy (Cb).
  * ρ is the Pearson correlation coefficient, which measures how far each observation deviates from the best-fit line, and is a measure of precision, and
  * Cb is a bias correction factor that measures how far the best-fit line deviates from the 45° line through the origin, and is a measure of accuracy.

SECONDARY OUTCOMES:
Means | Through study completion, an average of 1 year.
  Means of cf-PWV, br-PWV, and e-PWV. Arithmetic mean: the arithmetic mean x ¯ x¯ is the sum of all observations divided by the number of observations n.

CONTACTS AND LOCATIONS:
Locations (1):
- CDC center, Uberaba, Minas Gerais, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Silva MA, Oliveira AP, Queiroz AC, Spaziani AO, Fernandes LA, De Oliveira KA, Lopes VDS, Landim MP, Cosenso-Martin LN, Vilela-Martin JF. Correlation between estimated pulse wave velocity values from two equations in healthy and under cardiovascular risk populations. PLoS One. 2024 Apr 9;19(4):e0298405. doi: 10.1371/journal.pone.0298405. eCollection 2024. PMID 38593112
- [Background] Stergiou GS, Palatini P, Parati G, O'Brien E, Januszewicz A, Lurbe E, Persu A, Mancia G, Kreutz R; European Society of Hypertension Council and the European Society of Hypertension Working Group on Blood Pressure Monitoring and Cardiovascular Variability. 2021 European Society of Hypertension practice guidelines for office and out-of-office blood pressure measurement. J Hypertens. 2021 Jul 1;39(7):1293-1302. doi: 10.1097/HJH.0000000000002843. No abstract available. PMID 33710173
- [Background] Van Bortel LM, Laurent S, Boutouyrie P, Chowienczyk P, Cruickshank JK, De Backer T, Filipovsky J, Huybrechts S, Mattace-Raso FU, Protogerou AD, Schillaci G, Segers P, Vermeersch S, Weber T; Artery Society; European Society of Hypertension Working Group on Vascular Structure and Function; European Network for Noninvasive Investigation of Large Arteries. Expert consensus document on the measurement of aortic stiffness in daily practice using carotid-femoral pulse wave velocity. J Hypertens. 2012 Mar;30(3):445-8. doi: 10.1097/HJH.0b013e32834fa8b0. PMID 22278144
- [Background] McEvoy JW, McCarthy CP, Bruno RM, Brouwers S, Canavan MD, Ceconi C, Christodorescu RM, Daskalopoulou SS, Ferro CJ, Gerdts E, Hanssen H, Harris J, Lauder L, McManus RJ, Molloy GJ, Rahimi K, Regitz-Zagrosek V, Rossi GP, Sandset EC, Scheenaerts B, Staessen JA, Uchmanowicz I, Volterrani M, Touyz RM; ESC Scientific Document Group. 2024 ESC Guidelines for the management of elevated blood pressure and hypertension. Eur Heart J. 2024 Oct 7;45(38):3912-4018. doi: 10.1093/eurheartj/ehae178. No abstract available. PMID 39210715
- [Background] Stamatelopoulos K, Georgiopoulos G, Baker KF, Tiseo G, Delialis D, Lazaridis C, Barbieri G, Masi S, Vlachogiannis NI, Sopova K, Mengozzi A, Ghiadoni L, Schim van der Loeff I, Hanrath AT, Ajdini B, Vlachopoulos C, Dimopoulos MA, Duncan CJA, Falcone M, Stellos K; Pisa COVID-19 Research Group; Newcastle COVID-19 Research Group. Estimated pulse wave velocity improves risk stratification for all-cause mortality in patients with COVID-19. Sci Rep. 2021 Oct 12;11(1):20239. doi: 10.1038/s41598-021-99050-0. PMID 34642385
- [Background] Greve SV, Blicher MK, Kruger R, Sehestedt T, Gram-Kampmann E, Rasmussen S, Vishram JK, Boutouyrie P, Laurent S, Olsen MH. Estimated carotid-femoral pulse wave velocity has similar predictive value as measured carotid-femoral pulse wave velocity. J Hypertens. 2016 Jul;34(7):1279-89. doi: 10.1097/HJH.0000000000000935. PMID 27088638
- [Background] Hametner B, Wassertheurer S, Mayer CC, Danninger K, Binder RK, Weber T. Aortic Pulse Wave Velocity Predicts Cardiovascular Events and Mortality in Patients Undergoing Coronary Angiography: A Comparison of Invasive Measurements and Noninvasive Estimates. Hypertension. 2021 Feb;77(2):571-581. doi: 10.1161/HYPERTENSIONAHA.120.15336. Epub 2021 Jan 4. PMID 33390046
- [Background] Reference Values for Arterial Stiffness' Collaboration. Determinants of pulse wave velocity in healthy people and in the presence of cardiovascular risk factors: 'establishing normal and reference values'. Eur Heart J. 2010 Oct;31(19):2338-50. doi: 10.1093/eurheartj/ehq165. Epub 2010 Jun 7. PMID 20530030
- [Background] Sarafidis PA, Loutradis C, Karpetas A, Tzanis G, Piperidou A, Koutroumpas G, Raptis V, Syrgkanis C, Liakopoulos V, Efstratiadis G, London G, Zoccali C. Ambulatory Pulse Wave Velocity Is a Stronger Predictor of Cardiovascular Events and All-Cause Mortality Than Office and Ambulatory Blood Pressure in Hemodialysis Patients. Hypertension. 2017 Jul;70(1):148-157. doi: 10.1161/HYPERTENSIONAHA.117.09023. Epub 2017 May 8. PMID 28483919
- [Background] Baumann M, Wassertheurer S, Suttmann Y, Burkhardt K, Heemann U. Aortic pulse wave velocity predicts mortality in chronic kidney disease stages 2-4. J Hypertens. 2014 Apr;32(4):899-903. doi: 10.1097/HJH.0000000000000113. PMID 24609217
- [Background] Salvi P, Scalise F, Rovina M, Moretti F, Salvi L, Grillo A, Gao L, Baldi C, Faini A, Furlanis G, Sorropago A, Millasseau SC, Sorropago G, Carretta R, Avolio AP, Parati G. Noninvasive Estimation of Aortic Stiffness Through Different Approaches. Hypertension. 2019 Jul;74(1):117-129. doi: 10.1161/HYPERTENSIONAHA.119.12853. Epub 2019 May 28. PMID 31132954
- [Background] Spronck B, Terentes-Printzios D, Avolio AP, Boutouyrie P, Guala A, Jeroncic A, Laurent S, Barbosa ECD, Baulmann J, Chen CH, Chirinos JA, Daskalopoulou SS, Hughes AD, Mahmud A, Mayer CC, Park JB, Pierce GL, Schutte AE, Urbina EM, Wilkinson IB, Segers P, Sharman JE, Tan I, Vlachopoulos C, Weber T, Bianchini E, Bruno RM; Association for Research into Arterial Structure and Physiology (ARTERY), the European Society of Hypertension Working Group on Large Arteries, European Cooperation in Science and Technology (COST) Action VascAgeNet, North American Artery Society, ARTERY LATAM, Pulse of Asia, and Society for Arterial Stiffness-Germany-Austria-Switzerland (DeGAG). 2024 Recommendations for Validation of Noninvasive Arterial Pulse Wave Velocity Measurement Devices. Hypertension. 2024 Jan;81(1):183-192. doi: 10.1161/HYPERTENSIONAHA.123.21618. Epub 2023 Nov 17. PMID 37975229
- [Background] Segers P, Rietzschel ER, Chirinos JA. How to Measure Arterial Stiffness in Humans. Arterioscler Thromb Vasc Biol. 2020 May;40(5):1034-1043. doi: 10.1161/ATVBAHA.119.313132. Epub 2019 Dec 26. PMID 31875700
- [Background] Townsend RR, Wilkinson IB, Schiffrin EL, Avolio AP, Chirinos JA, Cockcroft JR, Heffernan KS, Lakatta EG, McEniery CM, Mitchell GF, Najjar SS, Nichols WW, Urbina EM, Weber T; American Heart Association Council on Hypertension. Recommendations for Improving and Standardizing Vascular Research on Arterial Stiffness: A Scientific Statement From the American Heart Association. Hypertension. 2015 Sep;66(3):698-722. doi: 10.1161/HYP.0000000000000033. Epub 2015 Jul 9. No abstract available. PMID 26160955
- [Background] Safar ME, Toto-Moukouo JJ, Bouthier JA, Asmar RE, Levenson JA, Simon AC, London GM. Arterial dynamics, cardiac hypertrophy, and antihypertensive treatment. Circulation. 1987 Jan;75(1 Pt 2):I156-61. PMID 2947747
- [Background] Ben-Shlomo Y, Spears M, Boustred C, May M, Anderson SG, Benjamin EJ, Boutouyrie P, Cameron J, Chen CH, Cruickshank JK, Hwang SJ, Lakatta EG, Laurent S, Maldonado J, Mitchell GF, Najjar SS, Newman AB, Ohishi M, Pannier B, Pereira T, Vasan RS, Shokawa T, Sutton-Tyrell K, Verbeke F, Wang KL, Webb DJ, Willum Hansen T, Zoungas S, McEniery CM, Cockcroft JR, Wilkinson IB. Aortic pulse wave velocity improves cardiovascular event prediction: an individual participant meta-analysis of prospective observational data from 17,635 subjects. J Am Coll Cardiol. 2014 Feb 25;63(7):636-646. doi: 10.1016/j.jacc.2013.09.063. Epub 2013 Nov 13. PMID 24239664
- [Background] Safar ME, Asmar R, Benetos A, Blacher J, Boutouyrie P, Lacolley P, Laurent S, London G, Pannier B, Protogerou A, Regnault V; French Study Group on Arterial Stiffness. Interaction Between Hypertension and Arterial Stiffness. Hypertension. 2018 Oct;72(4):796-805. doi: 10.1161/HYPERTENSIONAHA.118.11212. No abstract available. PMID 30354723
- [Background] Lewington S, Clarke R, Qizilbash N, Peto R, Collins R; Prospective Studies Collaboration. Age-specific relevance of usual blood pressure to vascular mortality: a meta-analysis of individual data for one million adults in 61 prospective studies. Lancet. 2002 Dec 14;360(9349):1903-13. doi: 10.1016/s0140-6736(02)11911-8. PMID 12493255
- [Background] Franklin SS, Gustin W 4th, Wong ND, Larson MG, Weber MA, Kannel WB, Levy D. Hemodynamic patterns of age-related changes in blood pressure. The Framingham Heart Study. Circulation. 1997 Jul 1;96(1):308-15. doi: 10.1161/01.cir.96.1.308. PMID 9236450
- [Background] Mills KT, Stefanescu A, He J. The global epidemiology of hypertension. Nat Rev Nephrol. 2020 Apr;16(4):223-237. doi: 10.1038/s41581-019-0244-2. Epub 2020 Feb 5. PMID 32024986
- See also: Plataforma Brasil CAAE number : 57703722.7.0000.5415 — https://plataformabrasil.saude.gov.br/visao/pesquisador/gerirPesquisa/gerirPesquisaAgrupador.jsf